CLINICAL TRIAL: NCT06968845
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability and Efficacy of Caveolin-1-Scaffolding-Protein-Derived Peptide (LTI-03) in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: A Phase 2 Study of LTI-03 in Patients With Idiopathic Pulmonary Fibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rein Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LTI-03-2001 (RENEW)
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Idiopathic Pulmonary Fibrosis; Antifibrotic; Interstitial Lung Disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — Dry Powder Inhalers

STUDY DESIGN:
Intervention Model Description: LTI-03 and placebo are provided in powder-filled capsules that participants will self- administer using an inhaler. Placebo capsules look like LTI-03 capsules but have no active ingredients. Approximately 120 participants will be randomly assigned in a blinded manner to one of study drug treatment groups below.
  * Low dose LTI-03 (N=40) 1 inhaled capsule twice a day
  * Low dose placebo (N=20) 1 inhaled capsule twice a day
  * High dose LTI-03 (N=40) 2 inhaled capsules twice a day
  * High dose placebo (N=20) 2 inhaled capsules twice a day
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sponsor (1 unmasked Sponsor representative) CRO (1 Biostats individual is unmasked)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- (1) 2.5 mg LTI-03 capsule BID (Experimental): Caveolin-1-Scaffolding-Protein-Derived Peptide
  Interventions: Drug: LTI-03; Device: Dry Powder Inhaler
- (2) 2.5 mg LTI-03 capsules BID (Experimental): Caveolin-1-Scaffolding-Protein-Derived Peptide
  Interventions: Drug: LTI-03; Device: Dry Powder Inhaler
- (1) Placebo capsule BID (Placebo Comparator): Lactose powder
  Interventions: Device: Dry Powder Inhaler; Drug: Placebo
- (2) Placebo capsules BID (Placebo Comparator): Lactose powder
  Interventions: Device: Dry Powder Inhaler; Drug: Placebo

INTERVENTIONS:
Drug: LTI-03 — Caveolin-1-Scaffolding-Protein-Derived Peptide
  Arms: (1) 2.5 mg LTI-03 capsule BID; (2) 2.5 mg LTI-03 capsules BID
Device: Dry Powder Inhaler — Plastiape Monodose RS01 Model 7
Drug: Placebo — Lactose powder
  Arms: (1) Placebo capsule BID; (2) Placebo capsules BID

SUMMARY:
Rationale: LTI-03 is an experimental medication breathed into the lungs using an inhaler. It is being studied for the treatment of Idiopathic Pulmonary Fibrosis (IPF). IPF is a progressive, fatal lung disease caused by the death of lung cells involved in oxygen uptake and by progressive fibrosis (scarring) of the lungs. As the disease progresses, patients experience loss of lung function and increased breathing problems. LTI-03 is hypothesized to treat IPF by protecting and restoring the function of the oxygen uptake cells and by controlling lung fibrosis which may result in improving lung scarring.

The purpose of this research is to evaluate LTI-03 including: its safety, whether it causes side effects, whether it improves lung scarring, and whether it improves IPF symptoms. LTI-03 will be compared to placebo in patients diagnosed with IPF within the last 5 years. Patients on a stable dose of nintedanib, pirfenidone, or nerandomilast (if available by prescription) may participate.

Trial Design: This is a Phase 2, randomized, double-blind, placebo-controlled, multi-center study that includes a 28-day Screening Period, a 24-week Treatment Period, and 4-week Follow-up Period.

Study Assessments: Up to 9 visits to the study clinic will be required.

Safety and tolerability will be evaluated with the following assessments: physical examination; collection of vital sign data (heart rate, blood pressure, respiratory rate and peripheral oxygen saturation [SpO2] via pulse oximetry); heart data collected by 12-lead electrocardiogram; and collection of blood samples for safety laboratory tests. In addition, participants will be asked about any adverse events (side effects) they have experienced between clinic visits, if they have changed any medications, and if they are able to properly use their study drug inhaler.

Participants will undergo a lung function test (spirometry) at every visit, which will be used to evaluate both safety and efficacy. Another test measuring the diffusion capacity of the lungs for carbon monoxide (DLCO) will be required at Screening only.

Blood samples will also be collected at each visit to measure disease biomarkers. At select visits patients will be asked to complete the Living with Pulmonary Fibrosis questionnaire to evaluate their IPF symptoms. Participants will also undergo a specialized lung scan (HRCT) at Baseline and at the End of Treatment to measure changes in lung fibrosis.

Interventions: LTI-03 and placebo are provided in powder-filled capsules that participants will self- administer using an inhaler. Placebo capsules look like LTI-03 capsules but have no active ingredients. Approximately 120 participants will be randomly assigned in a blinded manner to one of study drug treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 40 years or older.
2. Willing and able to provide written informed consent.
3. Diagnosis of IPF within 5 years of Screening as confirmed by a centrally read HRCT of the chest as defined by the ATS/ERS/JRS/ALAT guideline. HRCT lung fibrosis by central read during screening must involve ≥ 10% of the lung and be greater than emphysema involvement of the lung.
4. Forced vital capacity (FVC) percent predicted ≥ 45% at Screening.
5. Diffusion capacity of the lungs for carbon monoxide (DLCO), hemoglobin-corrected percent predicted ≥ 30% within 8 weeks prior to Randomization.
6. Participants receiving nintedanib, pirfenidone, or nerandomilast (where approved for marketing) for IPF treatment must have been on a stable prescribed dose for at least 12 weeks prior to Randomization.
7. Participants who previously received nintedanib, pirfenidone, or nerandomilast must have discontinued treatment at least 8 weeks prior to Randomization.
8. Able to adequately self-administer study drug using the protocol-specified inhaler device.

Exclusion Criteria:

1. Forced expiratory volume in 1 second (FEV1)/FVC < 0.7 at Screening.
2. Use of N-acetyl cysteine or other supplements including but not limited to quercetin, omega-3 fatty acids, dehydroepiandrosterone, polyphenols, and phytochemicals within 7 days prior to Randomization and through Week 24.
3. Use of systemic corticosteroids at doses > 10 mg/day of prednisone or equivalent within 28 days prior to Randomization.
4. Active smoker.
5. Pulmonary exacerbation within 3 months prior to Screening.
6. Febrile pulmonary illness requiring antibiotic treatment within 28 days prior to Randomization.
7. Participation in a clinical study or treatment with an investigational drug or device within 28 days of the Screening Visit (or 5 half-lives of the investigational agent, whichever is longer).
8. History or evidence at Screening of significant renal impairment with estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2.
9. History or evidence at Screening of significant hepatic impairment with bilirubin > 3 mg/dL (> 51.3 μmol/L) and albumin < 2.8 g/dL (<28 g/L) and PT prolongation > 6 sec or INR > 2.3 while not on anticoagulant medication.
10. Active or history of malignancies within 5 years prior to Randomization, with the exception of localized nonmetastatic basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix, or prostate cancer.
11. Serious or active medical or psychiatric condition which, in the opinion of the Investigator, may interfere with treatment, assessment, or compliance with the protocol; or an expected survival of less than 24 weeks.

    Contraception and Pregnancy
12. Positive pregnancy test in female participants of childbearing potential (defined below).
13. Female participants who are lactating.
14. Females of childbearing potential (FOCBP) and men with partners of childbearing potential who do not agree to use an acceptable form of contraception for the duration of study treatment and for at least 90 days after the last dose of study drug. Male participants who do not agree to refrain from donating sperm during this same period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability as measured by the incidence of treatment-emergent adverse events (TEAEs) | Day 1 through Week 24

SECONDARY OUTCOMES:
Change from baseline in forced vital capacity (FVC) | Day 1 through Week 24
Change from baseline in percent predicted FVC | Day 1 through Week 24
Change from baseline in lung fibrosis measured by high resolution computed tomography (HRCT) | Day 1 through Week 24

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UAB Lung Health Center, Birmingham, Alabama
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - El Paso Pulmonary Association, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No